CLINICAL TRIAL: NCT06075732
Title: Academic-Community Team for Improving Vaccine Acceptability and Targeted Engagement: Public Housing
Brief Title: ACTIVATE in Public Housing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: vaccpublichousing
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Pneumonia; Influenza; Varicella Zoster; Meningitis; COVID-19; Vaccine Hesitancy
MeSH Terms: conditions — Pneumonia; Influenza, Human; Meningitis; COVID-19; Vaccination Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACTIVATE Leaders (Experimental): This is a one group pretest-posttest design to increase COVID-19 vaccine uptake and completion among African American and Latinx public housing residents in South Los Angeles. The proposed intervention will employ (1) culturally sensitive, (2) theoretically based intervention that will be jointly delivered by ACTIVATE triad leaders and researchers. The investigators will use the Information, Motivation, and Behavioral Skills (IMB) model and the Transtheoretical Model to implement the intervention. PRISM, a Dissemination and implementation (D&I) D&I-based model can guide the implementation of the ACTIVATE program for successfully expansion and maintenance in community settings, especially for under-resourced populations.
  Interventions: Behavioral: Increasing Willingness and Uptake of Influenza, Pneumonia, Meningitis, HZV, and COVID-19 Vaccination

INTERVENTIONS:
Behavioral: Increasing Willingness and Uptake of Influenza, Pneumonia, Meningitis, HZV, and COVID-19 Vaccination — Provide/enhance knowledge, modify attitudes, motivate and provide skills and resources to reduce Influenza, Pneumonia, Meningitis, HZV, and COVID-19 vaccine hesitancy and increase willingness and uptake in Influenza, Pneumonia, Meningitis, HZV, and COVID-19 vaccination.

SUMMARY:
This multilevel, multidisciplinary, theoretically based, culturally sensitive, community-engaged intervention sets out to mitigate uptake barriers and non-adherence to vaccination schedules as recommended by the CDC and increase influenza, meningitis, pneumonia, VZV, and COVID-19 vaccine rates among under-resourced African American and Latino public housing residents in South Los Angeles.

DETAILED DESCRIPTION:
Vaccinations are critical for preventing infectious diseases such as influenza, meningitis, pneumonia, varicella zoster virus (VZV), and COVID-19. Despite increasing national distribution and promotion of routine recommendations for adult vaccination, coverage remains low, with historically lower uptake among racial and ethnic minorities. This is compounded by higher levels of vaccine hesitancy, which may be attributed to a myriad of issues, including worsening social determinants, medical mistrust, and lack of access to health services. Specifically, African American and Latino public housing residents may benefit from public health campaigns and vaccination initiatives to support high vaccine uptake and confidence. This R01 proposal seeks to expand on a proven, multilevel, multidisciplinary, theoretically based, culturally sensitive, community-engaged intervention by expanding the Academic-Community Team for Improving Vaccine Acceptability and Targeted Engagement (ACTIVATE) program. Guided by a fusion of the Social-Ecological framework (SEM) and the Practical, Robust Implementation and Sustainability Model (PRISM), the ACTIVATE program is inclusive of health factors on the individual, interpersonal, community, and societal level and elements for successful implementation. Led by leadership triads of public housing resident leaders, nurse practitioner students, and public health students, the ACTIVATE program centers on mitigating uptake barriers and non-adherence to vaccination schedules as recommended by the CDC and to increase influenza, meningitis, pneumonia, VZV, and COVID-19 vaccine rates among under-resourced AA and Latino adults in South LA.

ELIGIBILITY:
Aim 3:

Inclusion Criteria:

* identify as Latinx or African American
* age 18 or older
* reside in one of the six collaborating public housing area
* Speak either English or Spanish
* Report vaccine hesitancy

Exclusion Criteria:

* Not a resident at one of the collaborating public housing areas
* Does not self-identify as African American or Latinx
* Age 17 and younger
* Unable to speak either English or Spanish
* Received all recommended vaccines for Influenza, Pneumonia, Meningitis, VZV, and COVID-19
* No reporting of vaccine hesitancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of vaccination uptake for Influenza, Pneumonia, Meningitis, VZV, and COVID-19 using Vaccination History Self Report | Intervention: 8 months; Follow-up Point: 3- and 9-months post-intervention
  By comparison of pre-, post- intervention, and 9- and 18-months follow-up data, the investigators anticipate the following compared to baseline: a 40% change in completion of Influenza, Pneumonia, Meningitis, VZV, and COVID-19 vaccination series

SECONDARY OUTCOMES:
Percentage of Participants Achieving Decreased Vaccine Hesitancy Levels of Influenza, Pneumonia, Meningitis, VZV, and COVID-19 vaccine Using the NIH Toolbox Surveys on COVID-19 | Intervention: 8 months; Follow-up Point: 3- and 9-months post-intervention
  By comparison of pre-, post- intervention, and 3- and 9-months follow-up data, the investigators anticipate the following compared to baseline: a 40% change in hesitancy toward Influenza, Pneumonia, Meningitis, VZV, and COVID-19 vaccination
Percentage of Participants Achieving Increased Level of Behavior Change toward COVID-19 Vaccination Using the NIH Toolbox Surveys on Influenza, Pneumonia, Meningitis, VZV, and COVID-19 | Intervention: 8 months; Follow-up Point: 3- and 9-months post-intervention
  By comparison of pre-, post- intervention, and 3- and 9-months follow-up data, the investigators anticipate the following compared to baseline: a 40% change in their behavior stage of change toward Influenza, Pneumonia, Meningitis, VZV, and COVID-19 vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Charles R. Drew University of Medicine & Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No